CLINICAL TRIAL: NCT06988332
Title: A Pilot, Single-blind, Randomized Controlled Trial Evaluating the Implementation Outcomes and Preliminary Efficacy of Problem Management Plus (PM+) Versus Treatment as Usual in Adult Primary Care Users With Symptoms of Depression and/or Anxiety
Brief Title: Problem Management Plus (PM+) in Chile: a Pilot Randomized Controlled Trial of a Psychological Transdiagnostic Intervention Delivered in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Pan American Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 390
Record Dates: First submitted 2025-04-24; First posted 2025-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorders; Depressive Disorder
Keywords: Common mental health disorders; Common mental health problems; Depressive disorder; Anxiety disorders; Pilot Randomised Controlled Trial; Pilot RCT; PM+; Problem Management Plus
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Management Plus (PM+) (Experimental): PM+ is delivered in five individual sessions conducted by trained healthcare professionals without previous expertise in mental health care.
  Interventions: Behavioral: Problem Management Plus (PM+)
- Care as Usual (CAU) (No Intervention): Care as usual comprises the mental health services currently provided to Primary Health Care users in Chile.

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — Problem Management Plus (PM+) will be delivered according to the Spanish version of the WHO protocol (OMS, 2016).
  PM+ is a low-intensity, transdiagnostic psychological intervention based on Cognitive Behavioral Therapy (CBT). The protocol incorporates evidence-based strategies, including problem-solving, stress management, behavioral activation, and accessing social support.
  The intervention consists of five individual 90-minute sessions provided by healthcare professionals without previous expertise in mental health care (WHO, 2018). PM+ helpers will be supervised by master trainers specifically trained for Chile.
  Two systematic reviews have demonstrated the effectiveness of PM+ in reducing symptoms of common mental disorders, such as depression and anxiety (Schäfer et al., 2023) and specific symptoms of post-traumatic stress (Akhtar et al., 2022).
  Arms: Problem Management Plus (PM+)

SUMMARY:
This study aims to evaluate the implementation outcomes of a pilot randomized controlled trial and to assess the preliminary efficacy of Problem Management Plus (PM+) in reducing symptoms of depression and anxiety among users at a Primary Health Care center in Chile.

Two intervention groups will be compared: PM+ versus care as usual (CAU). The process will include an evaluation of the feasibility of the study procedures, as well as the acceptability and fidelity of the PM+ intervention.

DETAILED DESCRIPTION:
In Chile, only 19% of the population with mental health conditions has access to primary care services, highlighting the urgent need to expand mental health care availability. Training more healthcare professionals to deliver low-intensity psychological interventions could be a valuable approach to addressing this disparity.

The World Health Organization's Problem Management Plus (PM+) is a low-intensity, transdiagnostic, peer-delivered intervention designed for implementation in resource-limited settings to address common mental health disorders. In this context, PM+ serves as an evidence-based strategy that can help reduce gaps in healthcare services, particularly regarding availability and accessibility.

This study aims to evaluate the implementation outcomes of a pilot randomized clinical trial, including feasibility, acceptability and fidelity and to assess the preliminary efficacy of PM+ in reducing mental health symptoms among users at a primary healthcare center in Chile.

The study design is a single-blind pilot randomized controlled trial with a 1:1 allocation ratio, assessing two intervention arms for participants with depressive and/or anxiety symptoms over five weeks.

The study population consists of adults of 18 years or above with mild to moderate depressive and/or anxiety symptoms, living in the selected study region and enrolled in the primary health care center chosen to conduct the trial.

Two groups will be compared. The treatment group will receive five sessions of PM+. The control group will receive care as usual (CAU), which includes the regular mental health services provided at the primary health care center selected for the study.

Implementation outcomes of PM+ will be assessed, focusing mainly on feasibility, acceptability and fidelity. Additionally, preliminary efficacy outcomes of depression, anxiety and self-identified problems will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years old.
* Diagnosed with or presenting depressive and/or anxiety symptoms (through screening).
* Residents of the selected study region.
* Part of the population enrolled and validated in the pilot primary health care facilities.

Exclusion Criteria:

* Suicidal risk requiring immediate or urgent referral to care services.
* Suffering from severe psychiatric disorders or substance use disorders.
* Being in situations of declared risk that require protection (e.g., domestic violence).
* Moderate or severe disability.
* Incapacitating medical illnesses.
* Receiving other mental health treatments that could lead to over-intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
Implementation outcome: Feasibility | Feasibility outcome component A will be collected once recruitment is completed. Component B will be collected at week 6, starting from the first intervention week.
  Measured through components A and B. A. Percentage of participant recruitment: defined as the proportion of participants who consented to enroll in the trial and were subsequently recruited.
  B. Participant adherence to PM+: defined as the average number of PM+ sessions attended by each participant.
Implementation outcome: Acceptability | Acceptability outcomes will be collected during the post-intervention assessment at week 6, starting from the first intervention week.
  Indicators of PM+ acceptability among users and trained facilitators, assessed with quantitative scales. For users, an adapted version of the Abbreviated Acceptability Rating Profile (AARP) will be administered. The AARP consists of 8 Likert-scale items, yielding total scores ranging from 8 to 48, with higher scores indicating greater acceptability. For facilitators, an adapted version of the Acceptability of Intervention Measure (AIM) will be used. The AIM comprises 5 Likert-scale items, producing scores ranging from 4 to 20, where higher scores reflect greater acceptability. For both measures, descriptive statistics will be reported using median and interquartile range (IQR), as well as mean and standard deviation (x̄ [SD]).
Implementation Outcome: Fidelity | Fidelity outcomes will be collected throughout the intervention period, from the first to the final intervention week (week 5).
  Indicators of PM+ fidelity will be assessed with a study-specific rubric developed based on expert judgement. The rubric consists of 5 items, each reflecting a component of proper PM+ delivery. Items range from 1 ("low fidelity") to 4 ("high fidelity"), with higher scores indicating greater fidelity. The reported statistics will include the median and interquartile range (IQR) for each item, and the mean and standard deviation (x̄ [SD]) for the overall fidelity score per assessed PM+ session.

SECONDARY OUTCOMES:
Preliminary pre-to-post effect of PM+ on depressive symptoms. | Measured through baseline at week 0 and post-intervention assessment at week 6, starting from the first intervention week.
  Measured using the Patient Health Questionnaire - 9 items (PHQ-9), with scores ranging from 0 to 27. Higher scores indicate increased symptom severity.
Preliminary pre-to-post effect of PM+ on anxiety symptoms. | Measured through baseline at week 0 and post-intervention assessment at week 6, starting from the first intervention week.
  Measured using the Generalized Anxiety Disorder - 7 item (GAD-7), with scores ranging from 0 to 21. Higher scores indicate increased symptom severity.
Preliminary pre-to-post effect of PM+ on self-identified problems. | Measured through baseline at week 0 and post-intervention assessment at week 6, starting from the first intervention week.
  Measured using the Psychological Outcome Profiles (PSYCHLOPS), with scores ranging from 0 to 20. Higher scores indicate increased self-identified problem severity.

CONTACTS AND LOCATIONS:
Overall Officials: Camila A. Solís, MSc., Study Chair — University of Chile
Locations (1):
- CESFAM Las Ánimas, Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will only be shared when required by regulatory institutions. In order to protect privacy and ensure the confidentiality of information, all data shared with research staff members without direct access to the case file will identify participants solely by their enrollment number and will be transmitted using depersonalized forms, such as the CRF. In the case it becomes necessary to share IPD with regulatory institutions, such as ethics committees or governmental agencies, the depersonalized enrollment number will be used to maintain the confidentiality of personal information.
  Personal information will only be shared with public health care services or as required under Chilean legislation.

REFERENCES:
- [Result] Schafer SK, Thomas LM, Lindner S, Lieb K. World Health Organization's low-intensity psychosocial interventions: a systematic review and meta-analysis of the effects of Problem Management Plus and Step-by-Step. World Psychiatry. 2023 Oct;22(3):449-462. doi: 10.1002/wps.21129. PMID 37713578
- [Result] Akhtar A, Koyiet P, Rahman A, Schafer A, Hamdani SU, Cuijpers P, Sijbrandij M, Bryant RA. Residual posttraumatic stress disorder symptoms after provision of brief behavioral intervention in low- and middle-income countries: An individual-patient data meta-analysis. Depress Anxiety. 2022 Jan;39(1):71-82. doi: 10.1002/da.23221. Epub 2021 Nov 9. PMID 34752690
- See also: Link to the Spanish version of the WHO Problem Management Plus (PM+) protocol. — https://iris.who.int/handle/10665/259696
- See also: Link to the English version of the WHO Problem Management Plus (PM+) protocol. — https://www.who.int/publications/i/item/WHO-MSD-MER-18.5